CLINICAL TRIAL: NCT03831126
Title: The Impact of Stress on Fetal Brain Development
Brief Title: Stress and Fetal Brain Development
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: PerFet_maternal_stress_fMEG
Record Dates: First submitted 2019-01-30; First posted 2019-02-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy
MeSH Terms: interventions — betamethasone sodium phosphate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- betamethasone treatment
  Interventions: Drug: Betamethason Sodium Phosphate

INTERVENTIONS:
Drug: Betamethason Sodium Phosphate — First measurement: 12-36 hours after betamethasone treatment Second measurement: within five days after betamethasone treatment and two weeks Third measurement (neonatal measurement): 1-8 weeks after birh

SUMMARY:
The current proposal aims to investigate the impact of acute stress on the fetal autonomic nervous system.

DETAILED DESCRIPTION:
Over the last decades there is growing evidence that increased maternal stress levels lead to an adverse effect on the physiological, metabolic and neuronal development of the fetus during gestation with possible long-lasting effects. Several studies showed that maternal stress also affects fetal endocrine processes during pregnancy and increases the risk for childhood and adult obesity. Thus, the aim of the study is to investigate the effect of acute stress related to the action of the artificial glucocorticoid betamethasone on fetal heart and brain activity. The fetal activity will be measured with biomagnetic sensors.

ELIGIBILITY:
Inclusion Criteria:

* German speakers (fluently)
* Gestational age between 28 and 34 weeks
* Treatment with Betamethasone for improvement of fetal lung function -

Exclusion Criteria:

* Smoking (regularly)
* Alcohol and drug consumption during pregnancy
* Congenital fetal disorders
* Women with bed rest
* acute depression or other psychiatric disorder (self report)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
fetal and maternal heart rate | 8 weeks
  Measurement by fMEG

SECONDARY OUTCOMES:
fetal and neonatal brain activity in response to auditory and visual stimuli | 8 weeks
  Measurement by fMEG

OTHER OUTCOMES:
blood sugar levels | 8 weeks
  Measurement by fMEG

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Department of Women's Health, Tübingen, Germany